CLINICAL TRIAL: NCT05219591
Title: Comparison of the Efficacy of Obstructive Sleep Apnea Treatment With CPAP With and Without the Use of Expiratory Pressure Relief Technology
Brief Title: Obstructive Sleep Apnea Treatment With CPAP With and Without the Use of Expiratory Pressure Relief Technology
Acronym: OSAEPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: expiratoryrelief
Record Dates: First submitted 2021-05-14; First posted 2022-02-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: The study will be carried out in 4 steps:
  1. During Polysomnography exam: Intermittent application of expiratory pressure relief (EPR), when the peak inspiratory flow will be measured with and without the application of EPR, on sleep stage called N2
  2. During Polysomnography exam: After the intermittent application of EPR, manual CPAP pressure titration will be performed with (CPAP-EPRon) and without EPR on (CPAP-EPRoff), under random order and a blinded observer.
  3. Use of outpatient CPAP, in random order, for a total of 3 weeks:
     i. adjusted to the previously titrated pressure CPAP-EPRoff, without the addition of EPR technology (1 week) and with the addition of EPR technology(1 week).
     ii. adjusted to the previously titrated pressure CPAP-EPRon, with the addition of EPR technology, for 1 week.
  4. Use of outpatient CPAP, in random order, for a total of 2 weeks:
     i. adjusted in automatic mode with adding EPR technology on (1 week) and off (1 week).
Who Masked: Participant, Investigator
Masking Description: Participant Masking: on steps 2, 3 and 4 Investigator Masking: on step 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polysomnographic night (Other): intermittent application of the EPR technology on CPAP device during step 2, on polysomnographic night of the study.
  Interventions: Device: EPR
- Outpatient CPAP use (Other): Application of EPR technology during outpatient CPAP usage, on steps 3 and 4 of the study
  Interventions: Device: EPR

INTERVENTIONS:
Device: EPR — application of EPR technology during CPAP treatment

SUMMARY:
Expiratory pressure relief (EPR) is a technology designed to improve patient comfort during continous positive airway pressure (CPAP) treatment for obstructive sleep apnea (OSA). The investigators hypothesized that the use of CPAP with EPR is less effective in controlling OSA when compared to CPAP without EPR, applied at the same treatment pressure. The investigators also hypothesized that the CPAP pressure necessary to abolish respiratory events during both manual and automatic CPAP titration with EPR will be greater than the pressure titrated with CPAP without EPR. OSA participants will undergo full polysomnography during CPAP and EPR will be turned on and off in order to test the impact of EPR on airflow and residual AHI.

DETAILED DESCRIPTION:
Participants will be recruited at the sleep clinic. The study will be carried out in 4 steps, the first 2 during one night of full polysomnography (PSG) and the last 2 during CPAP treatment for 4 weeks at home:

1) PSG part 1: Intermittent application of expiratory pressure relief (EPR) during inspiratory flow limitation. Peak inspiratory flow will be measured with and without turning EPR technology on. 2) PSG part 2: After the intermittent application of EPR, polysomnography with manual CPAP titration will be performed with EPR technology on (CPAP-EPRon) and without EPR (CPAP-EPRoff), under random order and one blinded observer.

3) CPAP: Use of outpatient CPAP, in random order, for a total of 3 weeks: i. adjusted to CPAP-EPRoff, without turning EPR on (1 week) and turning EPR on(1 week).

ii. adjusted to CPAP-EPRon, turning EPR on, for 1 week. 4) Use of outpatient CPAP, in random order, for a total of 2 weeks: i. adjusted in automatic mode without turning EPR on (1 week) and turning EPR on (1 week).

Before the start of step 1, participants will be assessed using questionnaires to assess excessive daytime sleepiness (Epworth Sleepiness Scale) and sleep quality (Pittsburgh Sleep Quality Index).

The investigators will perform physical examination with measurement of cervical and abdominal circumference, measurement of height, weight and blood pressure. The investigators will inspect the oropharynx and classify according to the modified Mallampati scale.

In steps 1 and 2 of the study, a CPAP device (model AirSense 10 AutoSet, ResMed Ltd.) will be used coupled to an adapted nasal mask (model ConfortGel Blue Nasal, Philips Respironics), with a sealed hole, which allows the passage of one pharyngeal intraluminal pressure catheter (Millar, Houston, TX, USA). In addition, a heated pneumotachograph (model 3700A, Hans Rudolf, Kansas City, MO) will be attached to the mask.

In steps 3 and 4 of the study, a CPAP device (model AirSense 10 AutoSet, ResMed Ltd.) will be used coupled to a nasal mask (model ConfortGel Blue Nasal, Philips Respironics). This equipment has a technology that allows to change the device settings remotely.

In all steps of the study, the expiratory pressure relief - EPR will be adjusted to level 3, corresponding to 3 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* aged eighteen or over
* already have baseline polysomnography showing a severe Apnea-Hypopnea Index (AIH), defined according to the current criteria of the American Academy of Sleep Medicine (AASM) as 30 events / hour of sleep or more
* already be using a continuous positive pressure device (CPAP) at a pressure equal to or greater than 9 cmH2O with good adherence, defined as an average use equal to or greater than 4 hours per day.

Exclusion Criteria:

Patients with:

* severe or decompensated respiratory or cardiac diseases
* previous pharyngeal surgery or other sleep disorders, such as parasomnias, narcolepsy or primary insomnia
* users of sedative medications such as opioids, benzodiazepines and muscle relaxants
* uncontrolled diabetes or hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Peak Inspiratory Flow | 1 day
  The value of the peak inspiratory flow, measured before and after the activation of expiratory pressure relief technology, on a flow limitation period of sleep
Titrated CPAP level | 1 day
  The titrated CPAP level with and without the application of expiratory pressure relief technology
Apnea and Hypopnea Index with CPAP on fixed mode | 15 days, 5 days each group
  The index of apnea and hypopnea measured with and without the expiratory pressure relief, measured with the titrated CPAP level, on fixed mode
Apnea and Hypopnea Index with CPAP on automatic mode | 14 days, 7 days each group
  The index of apnea and hypopnea measured with and without the expiratory pressure relief, with the titrated CPAP level, on automatic mode

SECONDARY OUTCOMES:
CPAP mask pressure | 1 day
  The level of the mask pressure with and without the application of the expiratory pressure relief technology, on the beginning of the inspiration
CPAP Leakage, with CPAP on fixed mode | 15 days, 5 days each group
  The leakage measured by the CPAP algorithm device, measured with and without the expiratory pressure relief technology, on the fixed titrated mode
CPAP Leakage, with CPAP on automatic mode | 14 days, 7 days each group
  The leakage measured by the CPAP algorithm device, measured with and without the expiratory pressure relief technology, on the automatic titrated mode
CPAP usage, with CPAP on fixed mode | 15 days, 5 days each group
  The amount of usage, per day, of the CPAP device, titrated on fixed mode, with and without the expiratory pressure relief technology
CPAP usage, with CPAP on automatic mode | 15 days, 5 days each group
  The amount of usage, per day, of the CPAP device, titrated on automatic mode, with and without the expiratory pressure relief technology

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil